CLINICAL TRIAL: NCT00862277
Title: Evaluation of the Persistence of Bactericidal Antibodies in Adolescents and Adults Who Received a Single Dose of Menactra® Four to Eight Years Earlier
Brief Title: Persistence of Bactericidal Antibodies in Adolescents and Adults Who Had Received a Single Dose of Menactra® Vaccine
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MTA64
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Meningococcal Infections; Meningitis
Keywords: Menactra®; Menomune®; Meningitis; Meningococcal Infections
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — Meningococcal Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Menactra® from Previous Studies: Subjects previously received only one dose of meningococcal vaccine, Menactra® in Study MTA04, MTA12, MTA19, or MTA21.
  Interventions: Biological: Menactra®
- Group 2: Menomune® from Previous Study: Subjects previously received only one dose of meningococcal vaccine, Menomune® in Study MTA04
  Interventions: Biological: Menomune®
- Group 3: Control: Meningococcal vaccine-naive age matched subjects

INTERVENTIONS:
Biological: Menactra® — 0.5 mL, Intramuscular (from a previous study)
  Groups: Group 1: Menactra® from Previous Studies
Biological: Menomune® — 0.5 mL, Intramuscular (from a previous study)
  Groups: Group 2: Menomune® from Previous Study

SUMMARY:
To evaluate the persistence of bactericidal antibodies in adolescents and adults who received one dose of Menactra® vaccine approximately four to eight years earlier

DETAILED DESCRIPTION:
Subjects who received one dose of Menactra® or Menomune® in study MTA04, MTA12, MTA19 (NCT00777790), or MTA21 (NCT00777257) will be eligible for enrollment in trial this study. All eligible subjects will provide a blood sample at Visit 1, after which their participation in the study will be terminated. An age-matched meningococcal-vaccine naïve control group will be recruited to provide a blood sample for baseline antibody level evaluation.

No vaccine will be administered in this study.

ELIGIBILITY:
Inclusion Criteria :

* For subjects aged ≥ 18 years: Informed consent form signed and dated by the subject
* For subjects aged < 18 years: Informed consent form signed and dated by the subject and the subject's parent/legal guardian
* Subject (and parent/legal guardian if subject is < 18 years of age) able to attend the scheduled visit and comply with all trial procedures
* For Group 1: Previously received only one dose of meningococcal vaccine (Menactra®, received in Study MTA04, MTA12, MTA19, or MTA21)
* For Group 2: Previously received only one dose of meningococcal vaccine (Menomune®, received in Study MTA04)
* For Group 3: Aged 14 through 27 years and never received any meningococcal vaccine

Exclusion Criteria :

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding inclusion
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroids therapy > 2 weeks
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the investigator
* Current alcohol abuse or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Receipt of blood or blood-derived products in the past 3 months that might interfere with the assessment of immune responses
* Known Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C seropositivity
* History of invasive meningococcal disease (confirmed either clinically, serologically, or microbiologically)
* For Groups 1 and 2: Previous vaccination (including booster) against meningococcal disease, with the exception of the Menactra® or Menomune® vaccination received in trial MTA04, MTA12, MTA19, or MTA21
* Subjects deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent
* Received oral or injected antibiotic therapy within the 72 hours prior to the blood draw (temporary criteria)

Ages: 14 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects that previously received only one dose of meningococcal vaccine, Menactra® in Study MTA04, MTA12, MTA19 (NCT00777790), or MTA21 (NCT00777257); or Menomune® in Study MTA04 and age-matched meningococcal vaccine-naive controls.
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (18):
- United States (18):
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Marietta, Georgia
  - Martinez, Georgia
  - Woodstock, Georgia
  - Bardstown, Kentucky
  - Omaha, Nebraska
  - Austintown, Ohio
  - Cleveland, Ohio
  - Erie, Pennsylvania
  - Greenville, Pennsylvania
  - Harleysville, Pennsylvania
  - Latrobe, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Wexford, Pennsylvania
  - Kingsport, Tennessee
  - Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 16 December 2008 to 16 March 2009 in 21 medical centers in the US.
Pre-assignment Details: A total of 763 participants who met the inclusion and exclusion criteria were enrolled. One participant withdrew before sampling and is excluded from analysis and this report.
Groups:
- Group 1: Menactra® From Previous Studies: Participants who previously received only 1 dose of meningococcal vaccine, Menactra®, in Study MTA04, MTA12, MTA19, or MTA21
- Group 2: Menomune® From Previous Study: Participants who previously received only one dose of meningococcal vaccine, Menomune®, in Study MTA04
- Group 3: Control: Meningococcal vaccine-naive, age-matched participants
Period: Overall Study
Arm/Group | Group 1: Menactra® From Previous Studies | Group 2: Menomune® From Previous Study | Group 3: Control
Started | 561 | 96 | 105
Completed | 560 | 94 | 100
Not Completed | 1 | 2 | 5
Not completed — Protocol Violation | 1 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Menactra® From Previous Studies | Group 2: Menomune® From Previous Study | Group 3: Control | Total
Number analyzed (Participants) | 561 | 96 | 105 | 762
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 205 | 0 | 57 | 262
  Between 18 and 65 years | 356 | 96 | 48 | 500
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.1 (2.87) | 23.3 (2.17) | 19.3 (3.98) | 19.7 (3.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 264 | 49 | 64 | 377
  Male | 297 | 47 | 41 | 385
Region of Enrollment [Number; unit: participants]
  United States | 561 | 96 | 105 | 762

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Bactericidal Antibody Titers for Meningococcal Serogroups A, C, Y, and W-135 at ≥ 8 and ≥ 128 at Enrollment
Time Frame: Day 0
Population: Serum Bactericidal Assay Baby Rabbit Complement antibody titers to each of the 4 meningococcal serogroups in the vaccine were evaluated in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Menactra® From Previous Studies | Group 2: Menomune® From Previous Study | Group 3: Control
Number analyzed (Participants) | 559 | 94 | 100
Percentage of Participants
  Serogroup A ≥ 8, [n = 557, 93, 99] | 53 | 34 | 20
  Serogroup A ≥ 128, [n = 557, 93, 99] | 50 | 29 | 17
  Serogroup C ≥ 8 [n = 557, 92, 99] | 39 | 28 | 16
  Serogroup C ≥ 128 [n = 557, 92, 99] | 31 | 22 | 12
  Serogroup Y ≥ 8 [n = 558, 93, 99] | 91 | 83 | 72
  Serogroup Y ≥ 128 [n = 558, 93, 99] | 85 | 77 | 62
  Serogroup W-135 ≥ 8 [n = 556, 92, 99] | 84 | 64 | 50
  Serogroup W-135 ≥128 [n = 556, 92, 99] | 77 | 55 | 47

2. Primary Outcome: Geometric Mean Titers of Serum Bactericidal Antibody Assay Using Baby Rabbit Complement (SBA-BR) at Enrollment
Time Frame: Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Menactra® From Previous Studies | Group 2: Menomune® From Previous Study | Group 3: Control
Number analyzed (Participants) | 559 | 94 | 100
Titers
  Serogroup A [n = 557, 93, 99] | 74.0 [58.2 to 94.2] | 19.1 [11.7 to 31.2] | 11.0 [7.08 to 17.0]
  Serogroup C [n = 557, 92, 99] | 24.9 [20.1 to 30.7] | 16.9 [9.91 to 28.7] | 8.58 [5.86 to 12.6]
  Serogroup Y [n=558, 93, 99] | 369 [317 to 430] | 183 [121 to 277] | 84.1 [54.9 to 129]
  Serogroup W-135 [n = 556, 92, 99] | 246 [205 to 295] | 59.4 [37.6 to 93.8] | 38.7 [23.6 to 63.3]

ADVERSE EVENTS:
Time Frame: There were no safety outcomes; safety data were not collected in this study.
Arm/Group | Group 1: Menactra® From Previous Studies | Group 2: Menomune® From Previous Study | Group 3: Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications